CLINICAL TRIAL: NCT06450574
Title: Prospective, Controlled and Randomized Phase III Multicentric Study of the Treatment of T1,N0,M0 Rectal Cancer. Neoadjuvant Therapy and Transanal Endoscopic Surgery vs. Transanal Endoscopic Surgery (TAUTEM-T1 Study)
Brief Title: Preoperative Chemoradiotherapy and Transanal Endoscopic Microsurgery Versus Ttransanal Endoscopic Microsurgery in T1 N0, M0 Rectal Cancer (TAUTEM-T1 Study)
Acronym: TAUTEM-T1
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Xavier Serra-Aracil, Associate Professor. Medical Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAUTEM-T1_2024-01
Record Dates: First submitted 2024-05-19; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-05

CONDITIONS: Rectal Cancer Stage I
Keywords: Preoperative chemoradiotherapy; Transanal endoscopic microsurgery; Rectal Cancer; T1-N0-M0 Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Transanal Endoscopic Microsurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemoradiotherapy+TEM (Experimental): Preoperative chemotherapy: capecitabine 825 mg/m2 every 12 hours orally, plus Radiotherapy (50.4 Gy). After 10 weeks, transanal endoscopic microsurgery (TEM) is done
  Interventions: Drug: Capecitabine (Xeloda); Radiation: 50.4 Gy; Procedure: Transanal Endoscopic Microsurgery (TEM)
- ransanal endoscopic microsurgery (TEM) (Active Comparator): Transanal endoscopic microsurgery (TEM)
  Interventions: Procedure: Transanal Endoscopic Microsurgery

INTERVENTIONS:
Drug: Capecitabine (Xeloda) — Capecitabine 825 mg/m2 every 12 hours orally on days of radiotherapy
  Arms: Chemoradiotherapy+TEM
Radiation: 50.4 Gy — Radiotherapy was administered in daily fractions of 1.8 Gy 5 days a week according to standard schema. The total dose is 45 Gy plus a boost of 5.4 Gy to the tumor area
  Arms: Chemoradiotherapy+TEM
Procedure: Transanal Endoscopic Microsurgery (TEM) — 10 weeks after Chemoradiotherapy
  Other Names: Transanal Endoscopic Operation (TEO); Transanal Minimal Invasive Surgery (TAMIS)
  Arms: Chemoradiotherapy+TEM
Procedure: Transanal Endoscopic Microsurgery — Standard surgical treatment of T1, N0, M0 rectal cancer. Early after diagnosis
  Other Names: Transanal Endoscopic Operation (TEO); Transanal Minimal Invasive Surgery (TAMIS)
  Arms: ransanal endoscopic microsurgery (TEM)

SUMMARY:
Introduction: The standard treatment for rectal adenocarcinoma is total mesorectal excision (TME), a technique involving resection of the rectum, with or without a temporary or permanent stoma. TME is associated with high morbidity and genitourinary alterations. On the other hand, transanal endoscopic surgery (TEM) allows access to tumors up to 20 cm from the anal margin, with much lower postoperative morbidity and without the need for ostomy. For T1, N0, M0 rectal adenocarcinomas without poor prognostic factors, TEM is the technique of choice. However, recent studies have described local recurrences of up to 20%. Our group, TAUTEM, has just completed a phase III clinical trial in T2-T3ab, N0, M0 rectal cancer, comparing preoperative chemoradiotherapy (CRT) and TEM versus TME, with very positive results in terms of postoperative morbidity, quality of life, and a local recurrence rate of 7.4%, not inferior to TME.

These results encourage our TAUTEM group to launch a similar project at the T1, N0, M0 stage, comparing standard TEM treatment versus QRT and TEM, aiming to improve rectal preservation outcomes and enhance results regarding local recurrence, distant recurrence, and oncologic survival.

Method: Prospective, controlled, randomized phase III multicenter clinical trial. Patients with rectal adenocarcinoma within 10 cm of the anal margin and up to 4 cm in size, staged as T1, N0, M0, will be included. These patients will be randomized into two groups: TEM after CRT and TEM alone. Postoperative morbidity and mortality, CRT side effects, and quality of life will be recorded. The minimum follow-up will evaluate rectal preservation and local recurrence and survival at two and three years. The sample size calculation for the study will be 106 patients.

Conclusions: The aim of the study is to improve oncological outcomes in stage T1, N0, M0 rectal cancer through preoperative chemoradiotherapy associated with local surgery (TEM).

ELIGIBILITY:
Inclusion Criteria:

* Indication by multidisciplinary committee of indication for local excision, according to ESMO and NCCN criteria.
* Rectal adenocarcinomas in the biopsy, located at a distance from the anal margin less than or equal to 10 cm measured by rigid rectoscopy at the time of ER.
* Preoperative staging by ER and pelvic MRI of T1,N0. In case of disparity, higher staging will be considered the definitive diagnosis. If it is greater than T1, it will be excluded.
* Tumors equal to or less than 4 cm in maximum diameter measured by MRI.
* ASA index equal to or less than III.
* Absence of distant metastases by abdominal CT and chest X-ray (if inconclusive, Thoracic CT)

Exclusion Criteria:

* Preoperative staging by EER or pelvic MRI higher than T1 or N0.
* Presence of distant metastases. Synchrony with other colorectal adenocarcinomas.
* Undifferentiated rectal adenocarcinomas or with the presence of poor prognostic factors in the preoperative biopsy (undifferentiated, venous, lymphatic or perineural infiltration, budding) .
* Patients with intolerance to preoperative chemotherapy or radiotherapy.
* Do not sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Rectal preservation in T1,N0,M0 rectal cancer | 2 years
  Number of patients where local surgery has been maintained after applying the protocol exit criteria.minimum follow-up of 2 years in both groups.
Total mesorectal excision in T1,N0,M0 rectal cancer | 2 years
  Number of patients with Total mesorectal Excision (TME) after applying the protocol exit criteria.minimum follow-up of 2 years in both groups.

SECONDARY OUTCOMES:
Analysis of tolerance and side effects of preoperative chemoradiotherapy (CRT). | 30 days after preoperative CRT
  NCI Common Terminology Criteria for Adverse Events v3.0 after chemoradiotherapy, is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.
Postoperative morbidity and mortality in both groups. | 30 days after surgery
  Postoperative (30 days post-surgery): nosocomial, surgical, and non-surgical postoperative complications; complications according to the Dindo-Clavien classification and the CCI (Comprehensive Complication Index); hospital stay.
The clinical and pathological response of patients undergoing CRT. | 30 days after surgery
  The presence of a correct histological response after chemoradiotherapy is determined by the pathology study of the tumor excised after TEM, in order to establish TRG1 in Bouzourene's classification
Quality of life one year after surgery. | One year after surgery
  Law anterior resection syndrom (LARS), Wexner incontinence scale, EORTC QLQ-C30, EORTC QLQ-CR29, and Karnofsky quality of life questionnaires. Before treatment and One year after surgery en both groups
Local recurrence in both groups | At two years
  Local recurrence defined as the presence of adenocarcinoma in the biopsy on the residual scar, anastomosis, or the defect area of the excised tumor.
3-year survival results in both groups, | Three years
  3-year survival results in both groups, reflected in overall survival, disease-free survival (DFS), distant recurrence (DR), and rectal cancer survival.

IPD SHARING:
Plan to Share IPD: Undecided
SAP, Study Protocol, Informed Consent Form (ICF)

REFERENCES:
- [Background] Serra-Aracil X, Pericay C, Badia-Closa J, Golda T, Biondo S, Hernandez P, Targarona E, Borda-Arrizabalaga N, Reina A, Delgado S, Vallribera F, Caro A, Gallego-Plazas J, Pascual M, Alvarez-Laso C, Guadalajara-Labajo HG, Mora-Lopez L. Short-term outcomes of chemoradiotherapy and local excision versus total mesorectal excision in T2-T3ab,N0,M0 rectal cancer: a multicentre randomised, controlled, phase III trial (the TAU-TEM study). Ann Oncol. 2023 Jan;34(1):78-90. doi: 10.1016/j.annonc.2022.09.160. Epub 2022 Oct 8. PMID 36220461
- [Background] Serra-Aracil X, Pericay C. Reply to the Letter to the Editor 'The role of chemoradiotherapy in organ preservation for rectal cancer' by L. Xie, Q. Chen, and J. Zhu. Ann Oncol. 2023 Apr;34(4):440-442. doi: 10.1016/j.annonc.2022.12.011. No abstract available. PMID 37061250
- [Background] Casalots A, Serra-Aracil X, Mora-Lopez L, Garcia-Nalda A, Pericay C, Ferreres JC, Navarro-Soto S. T1 Rectal Adenocarcinoma: a Different Way to Measure Tumoral Invasion Based on the Healthy Residual Submucosa with Its Prognosis and Therapeutic Implications. J Gastrointest Surg. 2021 Oct;25(10):2660-2667. doi: 10.1007/s11605-021-04948-9. Epub 2021 Feb 24. PMID 33629231
- [Result] Serra-Aracil X, Pericay C, Golda T, Mora L, Targarona E, Delgado S, Reina A, Vallribera F, Enriquez-Navascues JM, Serra-Pla S, Garcia-Pacheco JC; TAU-TEM study group. Non-inferiority multicenter prospective randomized controlled study of rectal cancer T2-T3s (superficial) N0, M0 undergoing neoadjuvant treatment and local excision (TEM) vs total mesorectal excision (TME). Int J Colorectal Dis. 2018 Feb;33(2):241-249. doi: 10.1007/s00384-017-2942-1. Epub 2017 Dec 12. PMID 29234923
- [Result] Naik DN, Kaneda T. Biosynthesis of branched long-chain fatty acids by species of Bacillus: relative activity of three alpha-keto acid substrates and factors affecting chain length. Can J Microbiol. 1974 Dec;20(12):1701-8. doi: 10.1139/m74-263. No abstract available. PMID 4155346